CLINICAL TRIAL: NCT01568190
Title: An Open Trial to Asses the Tolerability of AVANZ Mite Mix Immunotherapy
Brief Title: An Open Trial to Assess the Tolerability of AVANZ Mite Mix Immunotherapy
Acronym: AV-M-01
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: ALK-Abelló A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-002017-11; 2011-002017-11 (EudraCT Number)
Record Dates: First submitted 2012-03-29; First posted 2012-04-02 (Estimated); Last update posted 2015-01-06 (Estimated); Status verified 2015-01

CONDITIONS: Allergic Rhinitis Due to Dust Mite
Keywords: House dust mites sensitisation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AVANZ (Experimental): AVANZ Mites
  Interventions: Biological: AVANZ MITE

INTERVENTIONS:
Biological: AVANZ MITE — Immunotherapy Dermatophagoides mix

SUMMARY:
The purpose of the trial is to assess the tolerability of the up-dosing phase of AVANZ Mite mix.

DETAILED DESCRIPTION:
The frequency of patients with adverse reactions will be the primary endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients 18-65 years of age.
* A clinical history of HDM induced allergic rhinoconjunctivitis with or without asthma at least one year prior to trial entry.
* Positive SPT to Dermatophagoides pteronyssinus (Der pte) or Dermatophagoides farinae (Der far) (wheal diameter ≥ 3 mm).
* A positive specific IgE against Der pte or Der far (≥Class 2; ≥0.70 KU/L) documenting in the last 5 years.

Exclusion Criteria:

* FEV1 < 70% of predicted value at screening after adequate pharmacologic treatment.
* Uncontrolled or severe asthma.
* A clinically relevant history of symptomatic perennial allergic rhinitis and/or conjunctivitis caused by an allergen, to which the subject is regularly exposed and sensitized.
* History of severe asthma exacerbation or emergency room visit or admission for asthma in the previous 12 months.
* At screening, current symptoms of, or treatment for, upper respiratory tract infection, acute sinusitis, acute otitis media or other relevant infection (serous otitis media is not an exclusion criterion).
* Treatment with parenteral corticosteroids, oral corticosteroids or anti-IgE in the previous 3 months or during the study (except for steroids if needed as rescue medication). Please, see Table 4.
* Currently treated with angiotensin converting enzyme (ACE) inhibitors, tricyclic antidepressants, β-blockers, mono amine oxidase inhibitors (MAOIs) and any other drug containing alum (e.g. antacids) taken on a daily basis.
* Previous treatment by other allergen concomitant IT or immunotherapy with HDM extracts within the previous 5 years (initiation of subcutaneous immunotherapy is acceptable if treatment has been discontinued before reaching maintenance dose; for SLIT 3 months in the last 5 years is accepted).
* History of anaphylactic shock due to e.g. food, insect venom, exercise or drug.
* History of severe and recurrent angioedema.
* Any contraindication according to the Investigator Brochure (IB).
* Use of an investigational drug within 30 days prior to screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2011-12; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Frequency of patients with adverse reactions. | Participants wil be followed for an expected average of 6 weeks.
  From date of inclusion until date of last visit documented, it's expected an average of 6 visits, assessed up to 6 weeks per subject.

SECONDARY OUTCOMES:
Frequency of patients with systemic reactions according to EAACI classification | Participants wil be followed for an expected average of 6 weeks.
  From date of inclusion until date of last visit documented, it's expected an average of 6 visits, assessed up to 6 weeks per subject.

CONTACTS AND LOCATIONS:
Overall Officials: ANA I TABAR, MD, Principal Investigator — HOSPITAL VIRGEN DEL CAMINO - PAMPLONA
Locations (1):
- Hospital Virgen Del Camino, Pamplona, Navarre, Spain

REFERENCES:
- [Derived] Tabar AI, Gonzalez Delgado P, Sanchez Hernandez C, Basagana Torrento M, Moreno Benitez F, Arina M. Phase II/III clinical trial to assess the tolerability and immunological effect of a new updosing phase of Dermatophagoides mix-based immunotherapy. J Investig Allergol Clin Immunol. 2015;25(1):40-6. PMID 25898693